CLINICAL TRIAL: NCT05302362
Title: Effect of Fixed vs. Tailored Intensity Transcranial Direct Current Stimulation for Attention Deficit After Traumatic Brain Injury: a Single Center, Prospective, Double Blind, Randomized-Controlled Clinical Trial, Pilot Study
Brief Title: Effect of Fixed vs. Tailored Intensity tDCS for Attention Deficit After TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TBI_tDCS
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2022-03

CONDITIONS: Traumatic Brain Injury; Attention Deficit; Cognitive Impairment
Keywords: traumatic brain injury; attention deficit; transcranial direct current stimulation
MeSH Terms: conditions — Brain Injuries, Traumatic; Attention Deficit Disorder with Hyperactivity; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Prospective, Double Blind, Randomized Controlled Clinical Trial ,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sham tDCS Group (Sham Comparator): Sham transcranial direct current stimulation using YMS-201B(YBrain, Daejeon, Korea); ramp-up 30sec to 1.5mA, 0mA stimulation for 19 min 30 sec.
  Interventions: Device: transcranial direct current stimulation
- Conventional tDCS Group (Active Comparator): Transcranial direct current stimulation using YMS-201B(YBrain, Daejeon, Korea); ramp-up 30sec to 1.5mA, continuous 1.5mA stimulation for 19 minutes, ramp-down 30sec to 0mA.
  Interventions: Device: transcranial direct current stimulation
- Tailored tDCS Group (Experimental): Transcranial direct current stimulation using YMS-201B(YBrain, Daejeon, Korea); ramp-up 30sec to 2.0mA, continuous 2.0mA stimulation for 19 minutes, ramp-down 30sec to 0mA.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Transcranial direct current stimulation using YMS-201B(YBrain, Daejeon, Korea)

SUMMARY:
Traumatic brain injury (TBI) is an important global health concern. Recently, advances in neurocritical care have led to an increase in the number of recovering TBI patients, and concomittantly in the incidence of complications of TBI. One of the most important sequalae of TBI is cognitive deficit, for which multimodal rehabilitation approach is indicated. Transcranial direct current stimulation (tDCS) is a promising treatment strategy for post-TBI cognitive deficits. However, a standardized tailored tDCS protocol is yet to be established for TBI patients. Therefore, this trial aims to 1) the efficacy of tDCS on post-TBI cognitive deficits, and 2) and optimized protocol of tDCS on post-TBI cognitive deficits via a three-arm double-blind, randomized controlled trial.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is an important global health concern. It is estimated that about 70 million individuals will suffer a traumatic brain injury (TBI) each year. Serious TBIs for hospitalization or death is at least 10 million annually. In 2006, Langlois et al reported that, 50,000 patients die directly from or complications related to TBI in the united states alone, and at least 5.3 million Americans suffer from long-term disabilities related to TBI.

Recently, advances in neurocritical care have led to an increase in the number of severe TBI patients recovering cognitive and physical function, eventually returning to independent life.

With the rising recovery rate of TBI patients, the number of complications of TBI is also rising. One of the most common sequalae of TBI is cognitive deficit. In 2004, Whiteneck et al reported that about 65% of patients who experienced moderate to severe TBI suffer from long-term cognitive deficit. Mild TBI patients show fewer and lighter symptoms of cognitive deficit. However, about 15% of patients suffer from persisting cognitive, emotional, behavioral, and physical disabilities after one year (Roe et al. Disabil Rehabil. 2009).

Common symptoms of post-TBI cognitive deficit are attention deficit, memory loss, and impaired cognitive proceessing (Salmond et al. Curr Opin Crit Care. 2005). Current treatment strategy of post-TBI cognitive rehabilitation constitute multimodal approach including "conventional" occupational therapy, computerized neurocognitive training (CNT), pharmacotherapy, and physical medicine.

Transcranial direct current stimulation (tDCS) is a treatment approach where direct current is applied transcranially, aiming to modulate local neuronal excitability. Previous researches have established that repeated tDCS is safe, cost-effective, and easily administered to various neurological disorders including TBI, stroke, Parkinsonism, Alzheimer's dementia, and multiple sclerosis.

Although cognitive improvements are reported, a standardized protocol of tDCS for TBI patients is yet to be established (Kang, J Korean Neurol Assoc. 2017). The repertoire of researches that studies the efficacy of tDCS on post-TBI cognitive deficits is limited, and further study is warranted to establish standardized protocol (Ulam et al. Clinical Neurophysiology 2015; Kang et al. Journal of Rehabilitation Medicine 2012; Sacco et al. Front. Behav. Neurosci. 2016; Lesiank et al. J Head Trauma Rehabil. 2014; Rushby et al. Neuropsych Rehabil 2020; Motes et al J. Neurotrauma 2020).

This trial aims to determine 1) the efficacy of tDCS on post-TBI cognitive deficits, and 2) and optimized protocol of tDCS on post-TBI cognitive deficits via a three-arm double-blind, randomized controlled trial. The hypotheses of this experiment are as follow:

1. Sham group and actual stimulation group will show significantly different aCPT response time after 10 tDCS sessions.
2. Within the actual stimulation group, tailored tDCS subgroup will show significantly better aCPT response time than conventional tDCS subgroup after 10 tDCS sessions.
3. Patients with EEG biomarker change will show significantly better aCPT response time than those without.

ELIGIBILITY:
Inclusion Criteria:

* 19 years or older
* At least 6 months since traumatic brain injury
* Cognitive disability measured by:

A) K-MoCA score 25 or below, or B) Trail making test A > 50.25s or B > 142.53s

Exclusion Criteria:

* Infection, open wound, bleeding, skull defect, or metal plates at or near tDCS site
* history of seizure
* Language disorder
* Serious cognitive deficit with K-MoCA score below 10
* Pregnancy or possibility of pregnancy
* MRI contraindications
* Previous medical history that may affect the patient's cognitive abilities (i.e. previous stroke, hypoxic ischemic encephalopathy, schizophrenia)
* Change in dosage of the following medications within the previous 2 weeks
* rivastigmine
* donepezil
* memantine
* antiepiletic medications

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Auditory Continuous Performance Test (aCPT) response time | 6 weeks
  The Auditory Continuous Performance Test (ACPT) screens for auditory attention deficits. In the test, patients are told that they will see or hear the numbers "1" or "2" and that they are to click the mouse when presented with a visual or auditory "1" and inhibit clicking when presented with a "2". The task is made more challenging by the shifting of modalities between the visual and auditory stimuli. Data are provided for over-all attentional functioning and response control, as well as separate visual and auditory attention and response control.

SECONDARY OUTCOMES:
Auditory Continuous Performance Test (aCPT) omission error, commission error | 6 weeks
  The Auditory Continuous Performance Test (ACPT) screens for auditory attention deficits. In the test, patients are told that they will see or hear the numbers "1" or "2" and that they are to click the mouse when presented with a visual or auditory "1" and inhibit clicking when presented with a "2". The task is made more challenging by the shifting of modalities between the visual and auditory stimuli. Data are provided for over-all attentional functioning and response control, as well as separate visual and auditory attention and response control.
Computerized Neurocognitive Test (CNT) | 6 weeks
  1. Digit span test: Digit span forward test follows the number played through the computer speaker as it is and a digit span backward test speaks in reverse.
  2. Verbal learning test: 15 target words are heard through the computer speaker, recalled in any order and the same target word is repeated five times. After listening to the target word five times, 15 new words are heard and then recalled for blocking and then the 15 target words are recalled again.
  3. Stroop test: 24 letters of "green," "blue," "yellow," and "red" and the corresponding colors are read as quickly as possible. Several tests consist of (A) reading black letters, (B) the test to read the color by presenting each color square, (C) the test to read letters that match the color of the letter, and (D) the test to read the color of the letter whose color that composes the letter does not match the letter. The response time is scored.
Cambridge Neuropsychological Test Automated Battery (CANTAB) | 6 weeks
  CANTAB tests changes in neuropsychological performance and include tests of working memory, learning and executive function; visual, verbal and episodic memory; attention, information processing and reaction time; social and emotion recognition, decision making and response control.
  1. Reaction Time (RTI) Reaction Time provides assessments of motor and mental response speeds, as well as measures of movement time, reaction time, response accuracy and impulsivity.
  2. Rapid Visual Information Processing (RVP) A white box is shown in the center of the screen, inside which digits appear in a pseudo-random order, at the rate of 100 digits per minute. Participants are requested to detect target sequences of digits When the participant sees the target sequence they must respond by selecting the button in the center of the screen as quickly as possible. The level of difficulty varies with either one- or three-target sequences that the participant must watch for at the same time.

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Mo Oh, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data can be shared on reasonable request

REFERENCES:
- [Background] Langlois JA, Rutland-Brown W, Wald MM. The epidemiology and impact of traumatic brain injury: a brief overview. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):375-8. doi: 10.1097/00001199-200609000-00001. PMID 16983222
- [Background] Kim HK, Leigh JH, Lee YS, Choi Y, Kim Y, Kim JE, Cho WS, Seo HG, Oh BM. Decreasing Incidence and Mortality in Traumatic Brain Injury in Korea, 2008-2017: A Population-Based Longitudinal Study. Int J Environ Res Public Health. 2020 Aug 26;17(17):6197. doi: 10.3390/ijerph17176197. PMID 32859061
- [Background] Whiteneck GG, Gerhart KA, Cusick CP. Identifying environmental factors that influence the outcomes of people with traumatic brain injury. J Head Trauma Rehabil. 2004 May-Jun;19(3):191-204. doi: 10.1097/00001199-200405000-00001. PMID 15247842
- [Background] Roe C, Sveen U, Alvsaker K, Bautz-Holter E. Post-concussion symptoms after mild traumatic brain injury: influence of demographic factors and injury severity in a 1-year cohort study. Disabil Rehabil. 2009;31(15):1235-43. doi: 10.1080/09638280802532720. PMID 19116810
- [Background] Salmond CH, Sahakian BJ. Cognitive outcome in traumatic brain injury survivors. Curr Opin Crit Care. 2005 Apr;11(2):111-6. doi: 10.1097/01.ccx.0000155358.31983.37. PMID 15758589
- [Background] Ferrucci R, Mameli F, Guidi I, Mrakic-Sposta S, Vergari M, Marceglia S, Cogiamanian F, Barbieri S, Scarpini E, Priori A. Transcranial direct current stimulation improves recognition memory in Alzheimer disease. Neurology. 2008 Aug 12;71(7):493-8. doi: 10.1212/01.wnl.0000317060.43722.a3. Epub 2008 Jun 4. PMID 18525028
- [Background] Cicerone KD, Goldin Y, Ganci K, Rosenbaum A, Wethe JV, Langenbahn DM, Malec JF, Bergquist TF, Kingsley K, Nagele D, Trexler L, Fraas M, Bogdanova Y, Harley JP. Evidence-Based Cognitive Rehabilitation: Systematic Review of the Literature From 2009 Through 2014. Arch Phys Med Rehabil. 2019 Aug;100(8):1515-1533. doi: 10.1016/j.apmr.2019.02.011. Epub 2019 Mar 26. PMID 30926291
- [Background] Boggio PS, Khoury LP, Martins DC, Martins OE, de Macedo EC, Fregni F. Temporal cortex direct current stimulation enhances performance on a visual recognition memory task in Alzheimer disease. J Neurol Neurosurg Psychiatry. 2009 Apr;80(4):444-7. doi: 10.1136/jnnp.2007.141853. Epub 2008 Oct 31. PMID 18977813
- [Background] Boggio PS, Ferrucci R, Mameli F, Martins D, Martins O, Vergari M, Tadini L, Scarpini E, Fregni F, Priori A. Prolonged visual memory enhancement after direct current stimulation in Alzheimer's disease. Brain Stimul. 2012 Jul;5(3):223-230. doi: 10.1016/j.brs.2011.06.006. Epub 2011 Jul 27. PMID 21840288
- [Background] Fregni F, Boggio PS, Santos MC, Lima M, Vieira AL, Rigonatti SP, Silva MT, Barbosa ER, Nitsche MA, Pascual-Leone A. Noninvasive cortical stimulation with transcranial direct current stimulation in Parkinson's disease. Mov Disord. 2006 Oct;21(10):1693-702. doi: 10.1002/mds.21012. PMID 16817194
- [Background] Boggio PS, Ferrucci R, Rigonatti SP, Covre P, Nitsche M, Pascual-Leone A, Fregni F. Effects of transcranial direct current stimulation on working memory in patients with Parkinson's disease. J Neurol Sci. 2006 Nov 1;249(1):31-8. doi: 10.1016/j.jns.2006.05.062. Epub 2006 Jul 14. PMID 16843494
- [Background] Benninger DH, Lomarev M, Lopez G, Wassermann EM, Li X, Considine E, Hallett M. Transcranial direct current stimulation for the treatment of Parkinson's disease. J Neurol Neurosurg Psychiatry. 2010 Oct;81(10):1105-11. doi: 10.1136/jnnp.2009.202556. PMID 20870863
- [Background] Fregni F, Thome-Souza S, Nitsche MA, Freedman SD, Valente KD, Pascual-Leone A. A controlled clinical trial of cathodal DC polarization in patients with refractory epilepsy. Epilepsia. 2006 Feb;47(2):335-42. doi: 10.1111/j.1528-1167.2006.00426.x. PMID 16499758
- [Background] Varga ET, Terney D, Atkins MD, Nikanorova M, Jeppesen DS, Uldall P, Hjalgrim H, Beniczky S. Transcranial direct current stimulation in refractory continuous spikes and waves during slow sleep: a controlled study. Epilepsy Res. 2011 Nov;97(1-2):142-5. doi: 10.1016/j.eplepsyres.2011.07.016. Epub 2011 Aug 31. PMID 21885255